CLINICAL TRIAL: NCT05259293
Title: Characteristics of Pneumothorax Associated With Transthoracic Percutaneous Lung Biopsy in Standard of Care: a Retrospective Study in 6 Centers
Brief Title: Characteristics of Pneumothorax Associated With Transthoracic Percutaneous Lung Biopsy in Standard of Care
Acronym: PNOrate
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021/625
Record Dates: First submitted 2021-12-07; First posted 2022-02-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-01

CONDITIONS: Pneumothorax Iatrogenic Postprocedural
Keywords: interventional radiology, iatrogenic pneumothorax, transthoracic lung biopsy, pneumothorax rate, pneumothorax characteristics, patient management

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention - retrospective study — This is a retrospective study. No intervention.

SUMMARY:
The number of lung biopsies has increased steadily in recent years. Pneumothorax is the most common complication of a lung biopsy and can occur during the procedure, immediately after the procedure or within a few hours (delayed pneumothorax). The incidence of pneumothorax in the literature is very different from one study to another: it has been reported to be from 9 to 54% in patients undergoing percutaneous transthoracic needle biopsy. This difference of incidence could be explained by the absence of consensus for the definition of an iatrogenic pneumothorax.

The characteristics of pneumothorax and the management of patients with iatrogenic pneumothorax will be evaluated in different centres in a retrospective manner. This study will contribute to refining the criteria for defining pneumothorax occurring during lung biopsy and will provide a better understanding of the condition and its management.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old and more at the time of the biopsy procedure in year 2020
* Having had a pneumothorax following their transthoracic percutaneous lung biopsy in year 2020

Exclusion Criteria:

* Objection to the use of the data (French sites only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who presented with a pneumothorax following their lung biopsy (see eligibility criteria)
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Annual incidence rate of pneumothorax related to transthoracic lung biopsy on total number of lung biopsies | 3 months

SECONDARY OUTCOMES:
Annual incidence rate of hospitalisation in patients with pneumothorax related to lung biopsies | 3 months
Annual incidence rate of drainage in patients with pneumothorax related to lung biopsies | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Julien BEHR, MD, Principal Investigator — CHU de Besançon
Locations (6):
- France (4):
  - CHU de Besançon, Besançon
  - Institut Bergonié, Bordeaux
  - CHU de Tours, Tours
  - Institut Gustave Roussy, Villejuif
- Saint James Hospital, Dublin, Ireland
- Oxford University Hospitals, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No